CLINICAL TRIAL: NCT05393466
Title: A Phase I/II, Open-label Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of BPI-361175 Tablets in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: BPI-361175 Tablets in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xcovery Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XCV-BPI361175-ONC-101
Record Dates: First submitted 2022-05-02; First posted 2022-05-26 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Non-small Cell Lung Carcinoma
Keywords: non-small cell lung carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase Ia Dose Escalation (Experimental): The number of patients enrolled will be determined based on the maximum number required to establish the RP2D according to a Bayesian Optimal Interval (BOIN) method and will depend on the true DLT rate. Up to 24 patients will be enrolled for the dose-finding part.
  Interventions: Drug: BPI-361175
- Phase Ib Expansion Study (Experimental): Based on clinical data obtained from Part 1a, up to 24 patients with advanced NSCLC harboring EGFR C797S mutation will be enrolled in this dose expansion part of the study. One or more dose levels may be investigated dependent on emerging data. The sample size will be determined based on practical considerations.
  Interventions: Drug: BPI-361175
- Phase II Study (Experimental): The phase II part will be conducted using a Bayesian Optimal Phase 2 (BOP2) method with efficacy monitoring based on cumulative information on Objective Response Rate (ORR). The BOP2 method will consist of 2 interim looks occurring when the number of evaluable patients reaches the pre-specified values of 10 and 20 and a final analysis when a total of 30 patients are evaluable.
  Interventions: Drug: BPI-361175

INTERVENTIONS:
Drug: BPI-361175 — BPI-361175 is an oral fourth-generation EGFR inhibitor. The activation of EGFR signaling pathways is associated with various biological events such as proliferation, migration, differentiation, and apoptosis.

SUMMARY:
This is a three-stage study, consisting of Phase Ia dose-escalation, Phase Ib dose expansion, and a Phase II component.

DETAILED DESCRIPTION:
This is a Phase I/II, open-label, non-randomized study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of BPI-361175 tablets in patients with advanced NSCLC with EGFR C797S mutation and other EGFR-related mutations. Adult patients (18 and above) will receive a single dose of BPI-361175 followed by a 7-day washout period with continuous oral dosing of BPI-361175 in 28 days cycle.

This is a three-stage study, consisting of Phase Ia dose-escalation, Phase Ib dose expansion, and pivotal Phase II study.

It is expected to provide a brand-new treatment for advanced NSCLC. The study design utilizes a Bayesian Optimal Interval (BOIN) method to guide the dose level assignment of BPI-361175 and estimate the MTD/RP2D based on cumulative information on DLTs in the Cycle 0 + Cycle 1 of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years old;
2. Life expectancy ≥ 12 weeks;
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
4. Patients with histologically or cytologically confirmed diagnosis of inoperable locally advanced or recurrent/metastatic NSCLC with EGFR mutations. Patients must have progressed from or be intolerant to or be unfit for standard treatment.
5. For dose escalation: patients with documented EGFR mutation that have progressed on or after third-generation EGFR-TKI. In addition, other lines of therapy may have been given.
6. For dose expansion and Phase II: patients with EGFR C797S mutation confirmed prior to enrollment on tissue or blood samples with radiological documentation of disease progression from first-generation, second-generation or third-generation EGFR-TKIs. In addition, other lines of therapy may have been given;
7. For dose expansion and Phase II, patients must have at least one measurable tumor lesion per RECIST v1.1 criteria as per Investigator's assessment;
8. Adequate bone marrow, liver, and renal function:

   * Blood: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (1500/mm3), platelets count ≥ 100 × 109/L, hemoglobin ≥ 9 g/dL (90 g/L) (must not have received transfusion or granulocyte colony-stimulating factor within 2 weeks of screening tests and procedures);
   * Liver function: total bilirubin ≤ 1.5 × ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 × ULN; if liver metastases exist, AST and ALT ≤ 5.0 × ULN; for patients with documented Gilbert's syndrome, total bilirubin ≤ 3.0 × ULN;
   * Renal function: Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min (calculated by CKD-EPI);
9. All acute toxic effects of any prior antitumor therapy or surgery must have resolved to baseline or ≤ CTCAE Grade 1 (with the exception of alopecia);
10. For women with childbearing potential, serum pregnancy test will be performed within 7 days before dosing, with a negative result, and they must be non-lactating; all patients should take medically recognized contraceptive measures throughout the treatment period and 3 months after the last dose (see section Error! Reference source not found.);
11. Men with partners of childbearing potential willing to use adequate contraceptive measures during the study and for 90 days after the last dose of study medication.
12. Patients must have fully understood and voluntarily signed informed consent form (ICF).

Exclusion Criteria:

1. Presence of another active primary malignant tumors;
2. Unstable, symptomatic primary CNS tumors/metastasis or leptomeningeal metastases which are not suitable for enrollment, as judged by investigators. A patient can be enrolled if his/her clinical condition is stable and imaging evidence does not show disease progression within 2 weeks prior to the first dose, and who is off corticosteroid, anticonvulsant or mannitol treatment for longer than 2 weeks prior to the first dose.
3. Treatment with the most recent therapy (e.g., chemotherapy, immunotherapy, targeted therapy, radiation therapy, investigational therapy/agent) within 4 weeks or approximately 5 half-lives, whichever is the longer, before the first dose. (If sufficient wash-out time has not occurred due to schedule or PK properties, an alternative appropriate wash-out time based on known duration and time to reversibility of drug related adverse events could be agreed upon by the sponsor and investigators);
4. Gastrointestinal disorders that would affect oral swallowing or the investigators judge the absorption of the study drug will be interfered;
5. Use of strong or moderate CYP3A inhibitors or inducers within 7 days prior to the first dose;
6. Autologous (within 3 months) or allogeneic (within 6 months) organ or stem cell transplantation prior to the first dose; any major surgery or severe trauma (except biopsy sampling) within 4 months prior to the first dose;
7. Palliative radiation therapy within 2 weeks prior to the first dose;
8. Patients who have active viral hepatitis B (HBV) infection (exception: HBV DNA ≤ 500 IU/mL and has been stable for longer than 4 weeks);
9. Patients who have active infections that required systemic therapy within 1 week prior to the first dose;
10. Any of the following cardiac conditions within the last 6 months:

    Unexplained or cardiovascular cause of presyncope or syncope, tachycardia, ventricular fibrillation, or sudden cardiac arrest. Prolonged corrected QT interval [mean resting corrected QT interval QTcF > 450 msec for males or > 470 msec for females from 3 electrocardiogram (ECG)];
11. Any > CTCAE Grade 1 prior to the first dose;
12. Medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease, any uncontrolled systemic disease, and other serious illnesses;
13. Patients with deep venous thrombosis, pulmonary embolism or any other serious thromboembolism within 3 months prior to the first dose (implantable venous access-port, catheter-related thrombosis or superficial venous thrombosis is not considered as "serious" thromboembolism);
14. The presence of drug abuse and medical, psychological, or social conditions that do not permit compliance with the protocol or will not be available for protocol-required study visits or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with adverse events and serious adverse events graded per National Cancer Institute Common Terminology Criteria for Adverse Events and dose limiting toxicities for BPI 361175 | 18 months
  To characterize the pharmacokinetics (PK) of BPI-361175 tablets in advanced NSCLC
Efficacy of BPI-361175 | 18 months
  To determine the recommended Phase II dose (RP2D).

SECONDARY OUTCOMES:
Tmax | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  Time to maximum plasma concentration
Tumor assessments | At the end of every even cycle
  RECIST
Determine maximum tolerated dose in milligrams of BPI-361175 | Baseline up to Completion of Cycle 1 (28 days)
  MTD
Cmax | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  maximum plasma concentration
AUC0-t | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  Area under the plasma concentration-time curve from zero to the time of the last measurable concentration, as calculated using the trapezoidal rule.
AUC0-∞ | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  Area under the plasma concentration-time curve from zero to infinity.
AUCextrap% | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  Percentage of the extrapolated area to the entire AUC.
λz | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  Terminal elimination rate constant, as obtained by log-linear regression of the terminal segment of the plasma concentration vs time curve.
t1/2 | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  Terminal half-life, as calculated based on formula t1/2 = Ln(2)/λz
Vz/F | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  Apparent volume of distribution, Vz/F = CL/F/λz.
CL/F | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  Apparent plasma clearance, CL/F = dose/AUC0-∞.
Tmax, ss | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  Time to maximum plasma concentration at steady state.
Cmax, ss | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  Maximum concentration at steady state.
Ctrough, ss | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  Trough concentration at steady state.
Cmin, ss | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  Minimum trough concentration at steady state.
Area under the plasma concentration-time curve from zero to the end of the dosing interval. | Baseline, Cycle 1 Day1, Day 8, Day 15, Day 22, Day 28, and Day 1 of additional cycles
  AUCss

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni C Selvaggi, MD, Study Director — Xcovery Holdings, Inc.

IPD SHARING:
Plan to Share IPD: No